CLINICAL TRIAL: NCT05088980
Title: A Multicenter, Evaluator-blinded, Randomized, No-treatment Controlled Study to Evaluate the Safety and Effectiveness of JUVÉDERM VOLBELLA With Lidocaine Injectable Gel for Correction of Infraorbital Hollowing in Chinese Population
Brief Title: Study to Assess Effectiveness and Adverse Events of JUVEDERM VOLBELLA With Lidocaine Injection in Correcting Infraorbital Hollowing in Chinese Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1932-702-008
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Infraorbital Hollowing
Keywords: Infraorbital Hollowing; JUVEDERM VOLBELLA With Lidocaine; Lidocaine; VOLBELLA with Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VOLBELLA with Lidocaine (Experimental): Participants will receive VOLBELLA with Lidocaine on Day 1 and followed for 12 months.
  Interventions: Device: VOLBELLA with Lidocaine
- Control Group (Placebo Comparator): Participants will be followed for 3 months. Participants can opt to receive VOLBELLA with Lidocaine after 3 months and followed for 9 months.
  Interventions: Device: VOLBELLA with Lidocaine

INTERVENTIONS:
Device: VOLBELLA with Lidocaine — Facial Injection
  Other Names: JUVEDERM VOLBELLA with Lidocaine

SUMMARY:
Aged appearance is often caused by an infraorbital hollowing, which is characterized as a sunken appearance of the eye that results in the casting of a dark shadow over the nasal lower eyelid, giving a fatigued appearance. This study will assess how safe and effective JUVEDERM VOLBELLA with Lidocaine is in correcting infraorbital hollowing in adult participants in China.

VOLBELLA with Lidocaine is an investigational product being developed for the correction of infraorbital hollowing. Participants are randomly assigned to 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 on 4 chance that participants will be assigned to control group. Around 160 adult participants seeking correction of infraorbital hollowing will be enrolled at approximately 8 sites across China.

Participants in treatment group will receive VOLBELLA with Lidocaine injections on Day 1 and followed for 12 months. Participants in control group are followed for 3 months. Participants in Control group can opt to receive VOLBELLA with Lidocaine injection after completion of 3 months and followed for 9 months.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants seeking improvement of infraorbital hollowing.
* Has Moderate or Severe infraorbital hollowing (grade 2 or 3 on the AIHS) for each eye as assessed by the evaluating investigator (i.e., both eyes must qualify but do not need to have the same score).
* Treating Investigator (TI) considers the participant's anatomy to be amenable to improvement to an Allergan Infraorbital Hollows Scale (AIHS) grade of 0 or 1 (None or Minimal).
* Participant must be in good health as determined by medical history, vital signs an TI's judgment, including no known active pandemic infection.
* Able, as assessed by the TI, and willing to follow study instructions (including compliance with the safety diary) and likely to complete all required study visits.
* Able to complete effectiveness self-assessments without the use of glasses (contact lens use is acceptable if they will be used for all participant self-assessments).

Exclusion Criteria:

* Has experienced trauma to the infraorbital area within 12 months before enrollment or has residual deficiencies, deformities, or scarring in the periorbital or cheek areas.
* Has active or recurrent inflammation or infection in either eye.
* Has active autoimmune disease.
* Has history of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid (HA) products, or Streptococcal protein.
* Has received botulinum toxin treatment above the subnasale within 9 months before enrollment.
* Has changes in use of over-the-counter or prescription oral or topical, anti-wrinkle products above the subnasale within 30 days before enrollment.
* Current enrollment in an investigational drug or device study or participation in such a study within 30 days of entry into this study.
* Has tattoos, piercings, or scars that would interfere with visual assessment of the infraorbital hollows.
* TI's discretion based on participant's safety and/or study integrity (the participant has a condition or is in a situation that, in the TI's opinion, may put the participant at significant risk, may confound the study results, or may interfere significantly with the participant's participation in the study, such as clinically significant abnormal lab testing results as judged by TI).
* Directly or indirectly involved in the conduct and administration of this study as an investigator, subinvestigator, study coordinator, or other study staff member; employee of the sponsor; first-degree family member, significant other, or relative residing with one of the above persons involved directly or indirectly in the study; or enrolled in the study at another clinical site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for Evaluating Investigator's (EI) live assessment of AIHS | Month 3
  A "responder" is a participant with at least 1- grade improvement on the Allergan Infraorbital Hollows Scale (AIHS) in both infraorbital areas. AIHS is a 5-point ordinal scale developed by Allergan to grade the severity of infraorbital hollowing (0 = None, 4 = Extreme).

SECONDARY OUTCOMES:
Percentage of Participants Achieving "Responder" Status for EI's Assessment of GAIS | Month 3
  A "responder" is a participant who shows improvement in the overall aesthetic assessment in the infraorbital area using Global Aesthetic Improvement Scale (GAIS).
Percentage of Participants Achieving "Responder" Status for Participant's Assessment of GAIS | Month 3
  A "responder" is a participant who shows improvement in the overall aesthetic assessment in the infraorbital area using Global Aesthetic Improvement Scale (GAIS).
Change From Baseline of Overall Score in Participant Responses to FACE-Q Appraisal of Lower Eyelids Questionnaire | Month 3
  In the FACE-Q Appraisal of Lower Eyelids questionnaire, the responses to the 7 items will be summed and converted to a Rasch-transformed score that ranges from 0 to 100.

CONTACTS AND LOCATIONS:
Overall Officials: ALLERGAN INC., Study Director — Allergan
Locations (7):
- China (7):
  - Beijing Hospital /ID# 227588, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital /ID# 227590, Beijing, Beijing Municipality
  - Peking University First Hospital /ID# 227593, Xicheng District, Beijing Municipality
  - Nanjing Drum Tower Hospital /ID# 241042, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 241040, Nanjing, Jiangsu
  - The Affiliated Hospital of Qingdao University /ID# 227592, Qingdao, Shandong
  - Huashan Hospital, Fudan University /ID# 227591, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvieclinicaltrials.com/study/?id=1932-702-008#additional-resources-section